CLINICAL TRIAL: NCT04877067
Title: Bioretina Inc Ankara University Technopolis
Brief Title: Therapy of Toxic Optic Neuropathy Via Combination of Stem Cells With Electromagnetic Stimulation
Acronym: Magnovision
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ankara Universitesi Teknokent (Other)
Collaborators: International Olympic Committee (Unknown)
Responsible Party: Principal Investigator, Umut Arslan, Principal Investigator, Ankara Universitesi Teknokent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56733164/203 E.1925
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Methanol Poisoning; Toxic Optic Neuropathy; Stem Cell Tyrosine Kinase 1 Y842X; Magnetic Field Exposure
Keywords: Toxic optic neuropathy; Wharton's jelly derived mesenchymal stem cell; Repetitive electromagnetic stimulation
MeSH Terms: conditions — Toxic Optic Neuropathy

STUDY DESIGN:
Intervention Model Description: The cases were divided into 3 groups according to their similar demographic characteristics. Prospective open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WJ-MSC combine witf rEMS (Active Comparator): WJ-MSC was applied first to the patients after necessary preparations. rEMS application was started 10 days after WJ-MSC application.
  Interventions: Biological: Wharton jelly derived mesenchymal stem cell; Device: Repetitive electromagnetic stimulation
- Only rEMS (Active Comparator): rEMS applications were repeated 10 times with a 1-week interval.
  Interventions: Device: Repetitive electromagnetic stimulation
- Only WJ-MSC (Active Comparator): WJ-MSC was applied only one time for both eyes.
  Interventions: Biological: Wharton jelly derived mesenchymal stem cell

INTERVENTIONS:
Biological: Wharton jelly derived mesenchymal stem cell — WJ-MSC
  Other Names: CordoSight
  Arms: Only WJ-MSC; WJ-MSC combine witf rEMS
Device: Repetitive electromagnetic stimulation — rEMS
  Other Names: Magnovision
  Arms: Only rEMS; WJ-MSC combine witf rEMS

SUMMARY:
The axons of the retinal ganglion cells combine to form the optic nerve. The optic nerve transmits electrical signals to the visual cortex by various synapses. Optic nerve axons are more sensitive to toxins than retina because they are outside the blood retinal barrier. Methanol, various solvents and heavy metals, carbon dioxide, antiarrhythmic, antiepileptic, antibiotics and some vasoactive drugs can cause toxic optic neuropathy. There is a different pathophysiology for each toxin. Methanol is easily accessible alcohol in all types of disinfectants. Methanol is converted into formaldehyde and formic acid while metabolized in the liver. Formaldehyde disrupts ATP synthesis by blocking mitochondrial function and oxidative phosphorylation. Formic acid causes demyelination as a result of metabolic acidosis. Neuroinflammation occurs when denatured proteins block axoplasmic flow. All these processes can lead to apoptosis and permanent vision loss. Sildenafil is a vasoactive drug used in erectile dysfunction. Sildenafil decreases optic nerve head blood flow. Neuroinflammation develops secondary to the cessation of axoplasmic flow after hypoxia. If hypoxia and neuroinflammatiom persists, apoptosis and permanent vision loss develop. Amiodarone is an ion channel blocker used in the treatment of cardiac arrhythmias. Long-term use may cause disruption of ion channel balance in the optic nerve. This condition leads to asymmetric neuroinflammation and apoptosis.

Wharton's jelly derived mesenchymal stem cells (WJ-MSC) can increase mitochondrial ATP synthesis with paracrine effects and suppress neuroinflammation with immunomodulatory effects. Repetitive electromagnetic stimulation (rEMS) can rearrange ion channel balances and axoplasmic flow. The aim of this prospective phase-3 clinical study is to investigate the effect of WJ-MSC and rEMS combination in the therapy of toxic optic neuropathies. This combination is the first study in the literature for the therapy of toxic optic neuropathies.

DETAILED DESCRIPTION:
This prospective, open-label clinical phase-3 study was conducted at Ankara University Faculty of Medicine, Department of Ophthalmology between April 2019 and April 2021. Thirty-six eyes of 18 patients with toxic optic neuropathy were included in the study. The primary toxic optic neuropathy (TON) diagnosis was made in emergency or intensive care clinics. Patients who admitted within 3 months after the first intervention were included in the study. All patients enrolled underwent a complete routine ophthalmic examination, including the best-corrected visual acuity (BCVA) measurement with the early treatment of diabetic retinopathy study (ETDRS) chart (Topcon CC 100 XP, Japan). The patients were further evaluated with optical coherence tomography angiography (OCTA) from RTVue XR (Avanti, Optovue, Fremont, CA, USA) to analyse and measure the changes in the ganglion cell complex (GCC) layer that provided a typical co-registered en-face and cross-sectional multimodal imaging platform. Functional evaluation of optic nerve was followed by Compass 24/2 visual field (VF) test (Compass, CenterVue, Padova, Italy) and 120' pattern visual evoked potential (pVEP) test (Mon 2018F, Metrovision, Perenchies, France).

Subjects Thirty-six eyes of 18 TON patients were included in the study.

Inclusion criteria consisted of several parameters:

* Cases poisoned with a toxic agent within 3 months
* Patients with BCVA better than 35 letters
* Any degree of visual field loss
* Patients over 18 years old

Exclusion criteria consisted of several parameters:

* Cases poisoned with a toxic agent more than 3 months
* Patients with BCVA less than 35 letters: to perform the visual field test correctly
* Neurological sequelae that cannot be cooperated
* Smoking

The same treatment protocol was applied to all patients with methanol intoxication before admission to our clinic. Hemodialysis, bicarbonate and ethanol were administered to all patients. The cases were divided into 3 groups according to similar demographic characteristics.

Group 1: Consists of 12 eyes of 12 patients treated with WJ-MSC and rEMS combination in one eye. WJ-MSC was applied only one time before rEMS applications. rEMS application was started 10 days after WJ-MSC application.The rEMS was applied with a custom-designed helmet for 30 minutes after the WJ-MSC application. rEMS applications were repeated 10 times with a 1-week interval. The course was evaluated by comparing the BCVA, FPDI, GCC thickness, pVEP-p100 latency and amplitude parameters before and 3rd month of aplications.

Group 2: Consists of 12 eyes of 12 patients treated with only rEMS in one eye. The rEMS was applied with a custom-designed helmet for 30 minutes. rEMS applications were repeated 10 times with a 1-week interval. The course was evaluated by comparing the BCVA, FPDI, GCC thickness, pVEP-p100 latency and amplitude parameters before and 3rd month of aplications.

Group 3: Consists of 12 eyes of 6 patients treated with only WJ-MSC in two eyes. WJ-MSC was applied only one time for both eyes. The course was evaluated by comparing the BCVA, FPDI, GCC thickness, pVEP-p100 latency and amplitude parameters before and 3rd month of aplications.

Umbilical cord Wharton's jelly-derived mesenchymal stem cells preparation The mesenchymal stem cells used in this study were isolated from Wharton's jelly of the umbilical cord that was collected allogenicly from a single donor with the mother's consent. The umbilical cord sample was treated following several steps. Briefly, cord tissue was washed twice with phosphate-buffered saline (Lonza, Switzerland) and the Wharton's jelly part was minced using forceps and a scalpel. Minced pieces were cultivated in a cell culture dish (Greiner Bio-One, Germany) with Dulbecco's modified Eagle's medium F12 (DMEM)-low glucose with no L-glutamine (Bilogical Industries, Israel) and 10% human AB serum (Capricorn, Germany), 1% 10.000 U/mL penicillin, and 10.000 μg/mL streptomycin (Gibco,USA). All cell preparations and cultivation procedures were conducted in a current Good Manufacturing Practice (cGMP) accredited laboratory (Onkim Stem Cell Technologies, Turkey). The culture-expanded cells were cryopreserved at P3 using standard cryopreservation protocols until used in the following experiment. CryoSure-DEX40 (WAK-Chemie Medical, Germany) containing 55% Dimethyl Sulfoxide and 5% Dextran 40 was used as cryopreservant. The cells were characterized at the time of cryopreservation using flow cytometric analysis to determine the expression of the positive cluster of differentiation (CD) surface markers, CD90, CD105, CD73, CD44, CD29, and negative for CD34, CD45, and CD11b. Using real-time polymerase chain reaction (qPCR), the expressions of several genes, such as tumor necrosis alpha (TNF alpha) and vimentin (VIM) were analyzed. Additionally, quality control analyses, such as mycoplasma and endotoxin analyses (using the PCR and LAL test combined with sterility analysis, respectively) were also completed. Cells were solubilized from cryopreservation before being prepared for injection. Average cell viability for each treatment was over 90.0%, and each patient received 2-6 x 106 cells in a 1.5 ml saline solution.

Injection of umbilical cord WJ-MSCs The WJ-MSCs suspension from the culture was delivered to the operating room by cold chain and used within 24 hours. A total of 1.5 ml of the WJ-MSC suspension was immediately injected into the subtenon space of each eye. The procedure was conducted under topical anesthesia with proparacaine hydrochloride drops (Alcaine, Alcon, USA) and sterile conditions. 5/0 atraumatic traction suture was applied to the limbus for easy access and manuplation to application area. Postoperatively, loteprednol and tobramycin combination eye drops were given four times per day for one week, and oral amoxicillin clavulonate (1 gr) was given twice a day for five days

Retinal repetitive electromagnetic stimulation (rEMS) The rEMS helmet (MagnovisionTM, Bioretina Biotechnology, Ankara, Turkey) stimulated the retina and visual pathways with an electromagnetic field strength of 2000 miligauss, frequency of 42 hertz, and duration 30 minutes. These values were previously determined to be effective for other clinical and preclinical studies.

Timeframe

The patients were evaluated at several study timepoints:

* T0 (baseline): immediately before the applications
* T1: 1rst month of applications
* T2: 3rd month of applications

Primary outcome measure • ETDRS visual acuity: The visual acuity scores obtained from the T0 and T2 examinations were analyzed and compared using statistical tests to determine effectiveness.

Secondary outcome measures

• Visual field sensitivity: Fundus perimetry deviation index (FPDI, %) FPDI was examined in the 24/2 visual field of the computerized perimetry records. The FPDI offers data explaining how many of the 100 flashing points and what percentage of the visual field could be correctly seen by the patient. For VF analysis, in order to avoid mistakes during the test, practice rounds were carried out three times before applications.

• Ganglion cell complex thickness (GCC thickness, µm): GCC is the thickness from the internal limiting membrane to the inner plexiform layer in the 3x3 mm of foveal area. The measurement done automatically by the OCTA device. GCC is the total thickness of the ganglion cells and retinal nerve fibers.

• Pattern visual evoked potential (pVEP) pVEP is a objective test that measures the electrical activity of the optical pathway in response to a light stimulus. The 120' patterns reveals responses from the all retinal quadrants. The measurements were taken according to the ISCEV standarts for both eyes. We used the 120'pattern VEP protocol, which combines p100 implicit time and amplitude, to create a numerical result.

ELIGIBILITY:
Inclusion Criteria:

* Cases poisoned with a toxic agent within 3 months
* Patients with BCVA better than 35 letters
* Any degree of visual field loss
* Patients over 18 years old

Exclusion Criteria:

* Cases poisoned with a toxic agent more than 3 months
* Patients with BCVA less than 35 letters: to perform the visual field test correctly
* Neurological sequelae that cannot be cooperated
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
ETDRS visual acuity: | Change from baseline BCVA at 3 months
  The visual acuity scores obtained from the T0 and T2 examinations were analyzed and compared using statistical tests to determine effectiveness.

SECONDARY OUTCOMES:
Visual field sensitivity: Fundus perimetry deviation index (FPDI, %) | Change from baseline FPDI at 3 months
  FPDI was examined in the 24/2 visual field of the computerized perimetry records. The FPDI offers data explaining how many of the 100 flashing points and what percentage of the visual field could be correctly seen by the patient. For VF analysis, in order to avoid mistakes during the test, practice rounds were carried out three times before applications.
Ganglion cell complex thickness (GCC thickness, µm): | Change from baseline GCC thickness at 3 months
  GCC is the thickness from the internal limiting membrane to the inner plexiform layer in the 3x3 mm of foveal area. The measurement done automatically by the OCTA device. GCC is the total thickness of the ganglion cells and retinal nerve fibers.
Pattern visual evoked potential (pVEP) | Change from baseline p100 latency and amolitude at 3 months
  pVEP is a objective test that measures the electrical activity of the optical pathway in response to a light stimulus. The 120' patterns reveals responses from the all retinal quadrants. The measurements were taken according to the ISCEV standarts for both eyes. We used the 120'pattern VEP protocol, which combines p100 implicit time and amplitude, to create a numerical result.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University Biotechnology Institute, Ankara, Türkiye
  - Umut Arslan, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly derived mesenchymal stem cells: preliminary clinical results. Stem Cell Res Ther. 2020 Jan 13;11(1):25. doi: 10.1186/s13287-020-1549-6. PMID 31931872
- [Background] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly-derived mesenchymal stem cells: prospective analysis of 1-year results. Stem Cell Res Ther. 2020 Aug 12;11(1):353. doi: 10.1186/s13287-020-01870-w. PMID 32787913
- [Background] Arslan U, Ozmert E. Treatment of resistant chronic central serous chorioretinopathy via platelet-rich plasma with electromagnetic stimulation. Regen Med. 2020 Aug;15(8):2001-2014. doi: 10.2217/rme-2020-0056. Epub 2020 Oct 27. PMID 33107400
- [Background] Ozmert E, Arslan U. Management of Deep Retinal Capillary Ischemia by Electromagnetic Stimulation and Platelet-Rich Plasma: Preliminary Clinical Results. Adv Ther. 2019 Sep;36(9):2273-2286. doi: 10.1007/s12325-019-01040-2. Epub 2019 Aug 5. PMID 31385285
- [Background] Arslan U, Ozmert E. Management of Retinitis Pigmentosa via Platelet-Rich Plasma or Combination with Electromagnetic Stimulation: Retrospective Analysis of 1-Year Results. Adv Ther. 2020 May;37(5):2390-2412. doi: 10.1007/s12325-020-01308-y. Epub 2020 Apr 18. PMID 32303913
- [Derived] Ozmert E, Arslan U. Management of toxic optic neuropathy via a combination of Wharton's jelly-derived mesenchymal stem cells with electromagnetic stimulation. Stem Cell Res Ther. 2021 Sep 27;12(1):518. doi: 10.1186/s13287-021-02577-2. PMID 34579767